CLINICAL TRIAL: NCT01300624
Title: Effect Of Verb Network Strengthening Treatment on Lexical Retrieval in Aphasia
Brief Title: Effect of Verb Network Strengthening Treatment (VNeST) on Lexical Retrieval in Aphasia
Acronym: VNeST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C7695-R
Record Dates: First submitted 2011-01-21; First posted 2011-02-21 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Aphasia
Keywords: Aphasia; therapy; treatment; verbs; sentences
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Verb Network Strengthening Treatment (Experimental): Verb Network Strengthening Treatment (VNeST) tasks involve the retrieval of nouns related to a target verb. For example, for the verb measure, participants would come up with people who measure and what they measure (e.g., carpenter/lumber, chef/sugar). They would then answer questions related to why, where, and when these things might occur (e.g., for carpenter/measure, they might say to get the right length of board, (why) at a construction site, (where) and when building a house (where). Cues and assistance are provided to the participants when they are unable to complete any given task. As the participants improve, cues are reduced.
  Interventions: Behavioral: Verb Network Strengthening Treatment

INTERVENTIONS:
Behavioral: Verb Network Strengthening Treatment — Treatment to improve word retrieval in sentences and discourse for persons with aphasia due to stroke.
  Other Names: aphasia treatment, anomia, sentence production, discourse

SUMMARY:
The purpose of this study is to evaluate the effect of Verb Network Strengthening Treatment (VNeST) on the ability to produce sentences and connected speech in persons with aphasia.

DETAILED DESCRIPTION:
Stroke is the leading cause of disability in the United States today, and aphasia, a language disorder that affects production and comprehension of language, remains one of the most devastating aspects of stroke recovery. The most prominent symptom of aphasia is difficulty retrieving words, especially in sentence production and connected speech (e.g., telling a story, having a conversation). The current project examines the effect Verb Network Strengthening Treatment (VNeST), a language therapy, on the ability of persons with moderate aphasia to retrieve words in sentences and connected speech. The primary goals of VNeST are to 1) increase the specificity of nouns and verbs in sentences, 2) maximize improvement to untrained words across a variety of language tasks, and 3) engage and challenge participants with salient and relevant treatment materials and activities. Persons with aphasia who are enrolled in the study will receive VNeST for 10 weeks for 4 hours per week. Treatment tasks involve the retrieval of nouns related to a target verb. For example, for the verb measure, participants would come up with people who measure and what they measure (e.g., carpenter/lumber, chef/sugar). They would then answer questions related to why, where, and when these things might occur (e.g., for carpenter/measure, they might say "to get the right length of board," (why) "at a construction site," (where) and "when building a house" (where)). Cues and assistance are provided to the participants when they are unable to complete any given task. As the participants improve, cues are reduced.

Prior to treatment, testing will be conducted on participants to establish their abilities to retrieve words in the following contexts: 1) naming pictures of objects and actions, 2) sentences, and 3) connected speech.

Participants and a family member or friend (i.e., proxy) will also complete a questionnaire about how the participant is able to communicate in everyday tasks (e.g., indicating yes or no, providing medical information).

During the treatment phase, sentence production abilities on items related to treatment will be examined in order to determine how word retrieval abilities are changing with treatment. After the completion of treatment, all measures examined prior to treatment (including the questionnaire) will be re-examined in order to determine whether improvement was observed. Additionally, participants will complete testing one more time 3 months after the completion of treatment to determine if post-treatment improvements were maintained.

Finally, an analysis of improvement over time across the treatment phase will be examined in order to determine the rate of improvement (or lack of it) over time. All statistical analyses will use group data (i.e., group design), but additional examination of improvements for each participant (i.e., single subject design) will also be conducted. Thus, the overall experimental design is a mix of group and single subject analyses. The findings from this study will help to inform aphasia treatment practices and potentially allow for a larger study with more participants in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with a diagnosis of aphasia
* primary language is English
* aphasia due to stroke

Exclusion Criteria:

* Functionally bilingual

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Edmonds, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Verb Network Strengthening Treatment: Treatment tasks involve the retrieval of nouns related to a target verb. For example, for the verb measure, participants would come up with people who measure and what they measure (e.g., carpenter/lumber, chef/sugar). They would then answer questions related to why, where, and when these things might occur (e.g., for carpenter/measure, they might say "to get the right length of board," (why) "at a construction site," (where) and "when building a house" (where). Cues and assistance are provided to the participants when they are unable to complete any given task. As the participants improve, cues are reduced.
Period: Overall Study
Arm/Group | Verb Network Strengthening Treatment
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of participants was based on pilot study results and consistent with the relevant literature.
Arm/Group | Verb Network Strengthening Treatment
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11
Noun naming [Mean (Standard Deviation); unit: Percentage of correct naming] — Participants were asked to name the 162 object pictures (e.g., basket, arm) from An Object and Action Naming Battery. There was no time limit, and their final response was scored. An average of their correct responses was then calculated.
  Percentage of correct naming | 79.9 (12.3)
Verb naming [Mean (Standard Deviation); unit: Percentage of correct naming] — Participants were asked to name the 100 action pictures (e.g., climbing, sitting) from An Object and Action Naming Battery. There was no time limit, and their final response was scored. An average of their correct responses was then calculated.
  Percentage of correct naming | 64.6 (18.2)
Trained sentence probes [Mean (Standard Deviation); unit: Percentage correct sentence production] — This task required the production of a sentence to a given picture (N=10). Each picture contained a person or animal doing something with/to something. E.g.,, "A carpenter is measures the lumber." For a sentence to be considered correct (1 point), it had to contain the correct subject (carpenter), verb (measure) and object (lumber). These words could not be substituted by pronouns (he) or general words (man). Articles and verb inflections (i.e., "the," "is," "ing") were not required.
  This task is called the "Trained Sentence Probes," because the verb was trained in treatment.
  Percentage correct sentence production | 20.4 (13.3)
Untrained sentence probe [Mean (Standard Deviation); unit: Percentage correct sentence production] — This task required the production of a sentence to a given picture (N=10). Each picture contained a person or animal doing something with/to something. E.g., "A farmer is weighing apples." To be correct (1 point), the sentence had to contain the correct subject (farmer), verb (weigh) and object (apples). These words could not be substituted by pronouns (he) or general words (man). Articles and verb inflections ("the," "is," "ing") were not required.
  This is called the "Untrained Sentence Probes," because the verb in the picture (weigh) was semantically related to a trained verb (measure).
  Percentage correct sentence production | 19.8 (11.0)
Complete Utterances in discourse [Mean (Standard Deviation); unit: Percentage of complete utterances] — We elicited 10 discourse responses that included personal information (What you do on Sundays), picture descriptions and procedural information (how to wash dishes) (Nicholas & Brookshire 1993). Each utterance was evaluated against the criteria for complete utterances (containing a subject, verb and object (if required) while ALSO being relevant). E.g., "The woman is something" lacks a main verb and is not fully informative, whereas "The woman is pouring a drink" is complete and relevant to the picture. Percentage of complete utterances relative to total number of utterances was calculated.
  Percentage of complete utterances | 39.7 (1.9)
Western Aphasia Battery [Mean (Standard Deviation); unit: units on a scale] — The Western Aphasia Battery-Revised is a standardized aphasia battery which evaluates the severity and type of aphasia. It is a criterion measure that results in an Aphasia Quotient (AQ) (range: 0-100, where lower scores indicate more severe aphasia). An AQ of 0-25 is very severe; an AQ of 26-50 is severe; an AQ of 51-75 is moderate; and AQ of 76 and above is mild. This aphasia quotient considers language production, comprehension and repetition. The score provided here is the mean AQ across participants.
  units on a scale | 75.9 (10.4)
Communicative Effectiveness Ratings [Mean (Standard Deviation); unit: units on a scale] — This questionnaire (Lomas et al, 1989) was provided to persons who communicated with the treatment participant regularly (e.g., a spouse). They rated how well the participant was able to perform on 16 common communication tasks (e.g., participating in a conversation over coffee). They rated each scenario along a line that spanned between the two extremes of ability, from "not at all able" to "as able as before the stroke." The line was 100 mm. To score responses, the place where they bisected the line was measured. An average of their responses across the 16 questions was calculated.
  units on a scale | 32.6 (65.3)

OUTCOME MEASURES:

1. Primary Outcome: Trained Sentence Probe
Description: Picture description task that include trained words.
Time Frame: pre-treatment, post-treatment and 3-months post-treatment (maintenance)
Measure: Mean (Standard Deviation); unit: percentage of correct sentences
Arm/Group | Verb Network Strengthening Treatment
Number analyzed (Participants) | 11
percentage of correct sentences
  Pre-treatment | 20.4 (13.3)
  Post-treatment | 58.8 (33.9)
  3 months post-treatment (maintenance) | 56.0 (29.9)

2. Primary Outcome: Untrained Sentence Probes
Description: Picture description with sentences containing untrained words.
Time Frame: pre-treatment, post-treatment and 3-months post-treatment (maintenance)
Measure: Mean (Standard Deviation); unit: percentage of correct sentences
Arm/Group | Verb Network Strengthening Treatment
Number analyzed (Participants) | 11
percentage of correct sentences
  Pre-treatment | 19.8 (11.0)
  Post-treatment | 40.9 (24.9)
  3 months post-treatment (maintenance) | 43.0 (27.5)

3. Secondary Outcome: Noun Naming
Description: Confrontation naming of 162 objects
Time Frame: pre-treatment and post-treatment
Measure: Mean (Standard Deviation); unit: percentage of correct naming
Arm/Group | Verb Network Strengthening Treatment
Number analyzed (Participants) | 11
percentage of correct naming
  Pre-treatment | 79.9 (12.3)
  Post-treatment | 85.1 (12.6)

4. Secondary Outcome: Verb Naming
Description: Confrontation of 100 action pictures
Time Frame: pre-treatment and post-treatment
Measure: Mean (Standard Deviation); unit: percentage of correct naming
Arm/Group | Verb Network Strengthening Treatment
Number analyzed (Participants) | 11
percentage of correct naming
  Pre-treatment | 64.6 (18.2)
  Post-treatment | 74.2 (16.0)

5. Primary Outcome: Complete Utterances in Discourse
Description: Sentence in discourse that were relevant to topic and syntactically correct
Time Frame: pre-treatment, post-treatment and 3-months post-treatment (maintenance)
Measure: Mean (Standard Deviation); unit: percentage of complete utterances
Arm/Group | Verb Network Strengthening Treatment
Number analyzed (Participants) | 11
percentage of complete utterances
  Pre-treatment | 39.7 (11.9)
  Post-treatment | 46.7 (16.0)
  3 months post-treatment (maintenance) | 47.9 (13.8)

6. Secondary Outcome: Western Aphasia Battery
Description: Standardized measure of aphasia severity
Time Frame: pre-treatment and post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verb Network Strengthening Treatment
Number analyzed (Participants) | 11
units on a scale
  Pre-treatment | 75.9 (10.4)
  Post-treatment | 82.1 (8.6)

7. Secondary Outcome: Communicative Effectiveness Ratings
Description: This questionnaire (Lomas et al, 1989) was provided to persons who communicated with the treatment participant regularly (e.g., a spouse). They rated how well the participant was able to perform on 16 common communication tasks (e.g., participating in a conversation over coffee). They rated each scenario along a line that spanned between the two extremes of ability, from "not at all able" to "as able as before the stroke." The line was 100 mm. To score responses, the place where they bisected the line was measured. An average of their responses across the 16 questions was calculated.
Time Frame: pre-treatment, post-treatment and 3-months post-treatment (maintenance)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Verb Network Strengthening Treatment
Number analyzed (Participants) | 9
units on a scale
  Pre-treatment | 32.6 (9.7)
  Post-treatment | 65.3 (11.2)
  3 months post-treatment (maintenance) | 58.3 (15.6)

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Arm/Group | Verb Network Strengthening Treatment
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes